CLINICAL TRIAL: NCT02997189
Title: A Multicenter, Randomized, Phase 2 Study to Assess the Feasibility, Safety and Efficacy of OTO-104 Given by Intratympanic Administration in Subjects at Risk for Ototoxicity From Cisplatin Chemotherapy Regimens in the Treatment of Cancer
Brief Title: Study of OTO-104 in Subjects at Risk From Cisplatin-Induced Hearing Loss
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Negative Efficacy Results from the recently completed Phase 3 study 104-201506
Sponsor: Otonomy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 104-201607
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Cisplatin Induced Hearing Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OTO-104 (Active Comparator): One of the subject's ears will receive up to three administrations of study drug prior to cisplatin-based therapy
  Interventions: Drug: OTO-104
- Control (No Intervention): The ear not receiving OTO-104 will receive no treatment

INTERVENTIONS:
Drug: OTO-104 — 12 mg dexamethasone administered intratympanically
  Arms: OTO-104

SUMMARY:
This is a multicenter, Phase 2 study to assess the feasibility, safety and efficacy of OTO-104 given by intratympanic administration in subjects at risk for ototoxicity from cisplatin chemotherapy regimens in the treatment of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged 6 months to 21 years inclusive.
* Subject is diagnosed with neuroblastoma, hepatoblastoma, osteosarcoma or extracranial germ cell tumors and has not been previously treated with cisplatin or carboplatin.
* Subject is scheduled to receive a chemotherapy regimen that includes a cumulative cisplatin dose of ≥ 200 mg/m2.
* Subject has normal baseline auditory function, defined as ≤ 20 dB from 2000 to 8000 Hz, in both ears and does not have a history of sensorineural hearing loss.

Exclusion Criteria:

* Subject has middle ear effusion upon clinical examination.
* Subject has a history of central nervous system radiotherapy that encompasses all or part of the cochlea or will receive such radiation therapy during the course of the study.
* Subject is receiving sodium-thiosulfate or amifostine therapy with chemotherapy.
* Subject is currently participating on a separate otoprotection clinical study.

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2017-09-26 (Actual); Study Completion 2017-09-26 (Actual)

PRIMARY OUTCOMES:
Feasibility assessed via a questionnaire | Up to 18 weeks
  Feasibility to assess incorporating OTO-104 with a cisplatin-based therapy regimen

SECONDARY OUTCOMES:
Hearing function in each ear according to SIOP-Boston Ototoxicity Scale | Up to 6 months
Safety as assessed by adverse events | Up to 6 months
Local tolerability as assessed by otoscopic examinations | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kathie Bishop, PhD, Study Chair — Otonomy, Inc.
Locations (1):
- Contact Otonomy call center for trial locations, San Diego, California, United States

REFERENCES:
- [Background] Fernandez R, Harrop-Jones A, Wang X, Dellamary L, LeBel C, Piu F. The Sustained-Exposure Dexamethasone Formulation OTO-104 Offers Effective Protection against Cisplatin-Induced Hearing Loss. Audiol Neurootol. 2016;21(1):22-9. doi: 10.1159/000441833. Epub 2016 Jan 21. PMID 26789647